CLINICAL TRIAL: NCT02483026
Title: Nutritional Deficiencies Preventive Treatment Prior to Laparoscopic Sleeve Gastrectomy: Controlled Clinical Study
Brief Title: Nutritional Deficiencies Preventive Treatment Prior to Laparoscopic Sleeve Gastrectomy
Acronym: LSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Ram Elazary, Head bariatric surgeon Hadassah Ein Cerem Medical Center, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LSGD1HMO-CTIL
Record Dates: First submitted 2015-04-18; First posted 2015-06-26 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Disorder of Bone Density and Structure, Unspecified; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Geritol; Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive supplements care pre-surgery (Experimental): Multi vitamins pills vitamin D
  Interventions: Dietary Supplement: Multi vitamin; Dietary Supplement: vitamin D
- Standard supplements care pre-surgery (Other): vitamin D (Vitamin D will be given in a reduced doses compared to the intervention group)
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: Multi vitamin — Multi vitamin
  Arms: Intensive supplements care pre-surgery
Dietary Supplement: vitamin D — Vitamin D

SUMMARY:
This study will examine the effect of providing a structured program of daily nutritional supplements for a 8 weeks of intervention prior to Sleeve Gastrectomy bariatric surgery on bone mass density status and formation of critical nutritional deficiencies years after the surgery.

DETAILED DESCRIPTION:
The present study hypothesis holds that providing an adequate nutritional supplements program prior to the surgery, combined with postoperative monitoring, will significantly lower the incidence of nutritional deficiencies in patients undergoing Sleeve Gastrectomy surgery, and will reduce complications arising from these pre-operative deficiencies.

The investigators plan to examine the effect of Vitamins supplementation prior to surgery on the status of postoperative deficiencies one year after the surgery. Evaluation of outcomes will be made based on the results of blood tests specified, and related tests of bone density.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for bariatric surgery
* BMI over 35 kg / m 2 accompanying morbidity or BMI over 40 kg / m 2,
* pre-operative evaluation standards with matching to carry sleeve gastrectomy surgery
* Vitamin D deficiency prior to surgery

Exclusion Criteria:

* patients who underwent bariatric surgery in the past
* psychiatric or mentally contraindication for the procedure
* lack of consent to follow-up
* endocrine problem that affects the weight that is unbalanced.
* Chronic kidney disease (CKD), nephrolithiasis
* Hypercalcaemia
* Hypercalciuria and renal stones nephrolithiasis
* Pregnancy, breastfeeding
* Using medications or disease condition known as affecting the status of calcium or bone metabolism 3 month prior to intervention
* Taking any nutritional supplements 2 weeks before the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
bone mass density | 1 year
  Status bone density one year after surgery will be measured by bone density test (DXA = X-ray dual energy absorptiometry) in units of g / cm2.

SECONDARY OUTCOMES:
Weight loss after the surgery | 1 year
  weight (kg), %excess weight loss ( %EWL).
Vitamin D status after the surgery | 1 year
  levels of vitamin D (ng/ml) and presence of vitamin D deficiency.
Vitamin B12 status after the surgery | 1 year
  levels of vitamin B12 (pg/dl) and presence of vitamin B12 deficiency.
Iron status after the surgery | 1 year
  levels of iron (µg/dl) and presence of iron deficiency.
Parathyroid hormone (PTH) status after the surgery | 1 year
  levels of Parathyroid hormone (PTH) (pg/ml)
Folate status after the surgery | 1 year
  levels of folate (ng/ml) and presence of folate deficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah hebrew university medical center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No